CLINICAL TRIAL: NCT06240871
Title: Contrast-enhanced Ultrasound and Non-invasive Pulmonary Artery Pressure Measurement
Brief Title: Contrast Enhanced PA Pressure Measurements
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Kameswari Maganti, Associate Professor, Northwestern University
Other Study IDs: STU00071358
Record Dates: First submitted 2014-12-08; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Pulmonary Hypertension
Keywords: Echo; PA pressures; comparison; Right Heart Catheterization
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pulmonary artery pressure measurements: The investigators will compare noninvasive right sided pressure measurements with invasive right heart catheterization performed in 3 steps:at rest, with agitated saline and with agitated echo contrast, Optison. This was not a clinical trial and there were no intervention arms per se. All patients received agitated saline and echocardiographic contrast.
  Interventions: Other: Pulmonary artery pressure measurements

INTERVENTIONS:
Other: Pulmonary artery pressure measurements — The investigators will compare noninvasive measurements of right sided pressure measurements with invasive RHC performed in 3 steps:at rest, with agitated saline and with agitated echo contrast, Optison. This was not a clinical trial and there were no intervention arms per se. All patients received agitated saline and echocardiographic contrast.

SUMMARY:
Pulmonary hypertension (PH) is an abnormal increase of the pressure inside the lung circulation. This condition can be caused by many different diseases. If PH persists for a long period of time, irreversible damage to the lung circulation and to the heart may ensue. A definitive diagnosis of PH requires direct measurement of the pressure within the lung circulation with a procedure called right heart catheterization (RHC). While overall safe, RHC is an invasive procedure and is associated with a small risk of complications (~1.1%) and, very rarely, death (0.055%), even when performed in experienced laboratories. Therefore, alternative diagnostic approaches are often employed such as an ultrasound technique called Doppler echocardiography which is non-invasive, relatively inexpensive and widely available technique. It is suitable not only as a screening tool but also for serial monitoring of disease progression in PH. However, the accuracy of Doppler echocardiography in measuring pressure in the lung circulation appears to be modest in patients with suspected PH. To improve the performance of Doppler echocardiography it is common practice to inject a small amount of agitated saline or an echocardiographic contrast medium (usually composed of microbubbles of fat containing a minuscule amount of a gas) into a vein. However, the accuracy of using agitated saline or a contrast agent in the measurement of pressures inside the lung circulation has not been established. The proposed study will assess the accuracy of Doppler echocardiographic measurements of pressures in the pulmonary circulation by simultaneously comparing the pressures collected during a RHC. The investigators will enroll 100 consecutive patients undergoing RHC in the Catheterization Laboratory of Northwestern Memorial Hospital. The investigators will measure pulmonary pressures by RHC and by Doppler echocardiography at baseline and following the injection of agitated saline as well as Optison®, an FDA-approved contrast agent commonly used in the echo laboratory. The investigators will then determine the accuracy of the Doppler echocardiography measurement without and with the use of agitated saline or Optison® with the measurements obtained during the RHC which is the gold standard. The results of this study will allow determination whether the use of echo contrast improves the accuracy of Doppler echocardiography and whether contrast-enhanced Doppler measurements are a clinically useful alternative to RHC measurements.

DETAILED DESCRIPTION:
Background Pulmonary hypertension (PH), defined as a mean pulmonary arterial pressure ≥ 25 mmHg at rest as assessed by right heart catheterization (RHC), is present in several clinical conditions1. While considered the gold standard for the measurement of pulmonary pressure, RHC is an invasive procedure and is associated with a small risk of morbidity (1.1%) and mortality (0.055%) even when performed at experienced centers2. Therefore, alternative diagnostic approaches are often employed. Doppler echocardiography is non-invasive, relatively inexpensive and widely available technique. It is potentially suitable not only as a screening tool for PH but also as a method for serial monitoring of disease progression. Among the echocardiographic methods introduced to indirectly measure pulmonary arterial pressure, the tricuspid valve regurgitant jet method and the pulmonary artery regurgitant jet method have been widely adopted3. By measuring with Doppler ultrasound the maximum velocity of the tricuspid regurgitant jet (v), the transtricuspid pressure gradient (Pg) can be calculated using the modified Bernoulli equation: Pg = 4v2. Right ventricular systolic pressure (RVSP) can then be estimated by adding the transtricuspid pressure gradient to the right atrial pressure (RAP), indirectly estimated by the diameter of the inferior vena cava (IVC) and the degree of its collapse during spontaneous respiration4. In the absence of pulmonary valve stenosis, the RVSP can be equated to the pulmonary arterial systolic pressure (PASP). Measurements of PASP by Doppler echocardiography show a very high correlation (r=0.93) with values obtained by RHC 5. However, the accuracy of Doppler echocardiography appears to be limited in the assessment of patients with suspected PH, in whom the difference in PASP determined by echo and by RHC may be overestimated or underestimated by greater than 10 mmHg6. To improve the performance of Doppler echocardiography, particularly in the presence of an inadequate jet of tricuspid regurgitation, it is common practice to use maneuvers such as the injection of agitated saline and/or echo contrast media such as Optison® (Perflutren Protein-Type A Microspheres Injectable Suspension, USP) to augment the tricuspid regurgitant velocity profile4. However, whether these maneuvers increase the accuracy of Doppler echocardiography in the assessment of right ventricular and pulmonary arterial pressures compared to standard Doppler echocardiography has not been investigated.

2. Research Methods Study Design Cross-sectional investigation to assess: 1) the correlations between right sided (right ventricular, pulmonary artery, and right atrial) pressures measured by RHC and by Doppler echocardiography in the absence of contrast and during the intravenous administration of agitated saline or Optison®; and 2) to compare such measures by assessment modality. The investigators hypothesize that the correlations between right sided pressures measured by Doppler echo during agitated saline or Optison® will be higher than those measured in the absence of a contrast agent, and that the correlations between right sided pressures measured by Doppler echo during Optison® will be higher than those measured during agitated saline.

The main correlations explored in the study will be:

Correlation between right atrial pressure measured by RHC and by Doppler echocardiography in the absence of a contrast agent.

Correlation between right ventricular pressure measured by RHC and by Doppler echocardiography in the absence of a contrast agent and during the intravenous administration of agitated saline or Optison®.

Correlation between PASP measured by RHC and by Doppler echocardiography in the absence of a contrast agent and during the intravenous administration of agitated saline or Optison®.

The main comparisons performed in the study will be:

Comparison between PASP measured by Doppler echocardiography in the absence of a contrast agent and the PASP measured during the intravenous administration of agitated saline or Optison®.

Comparison between PASP measured by Doppler echocardiography during the intravenous administration of agitated saline and during the intravenous administration of Optison®.

Study Population This study will include unselected consecutively patients 18 to 80 years old referred for RHC to the Cardiac Catheterization Laboratory of Northwestern Memorial Hospital. The informed consent for RHC will be obtained as part of the clinical assessment. A study physician will then approach patients and eligibility will be assessed. A separate informed consent will be obtained for the limited Doppler echocardiographic study to be performed simultaneously during the RHC in patients interested in participating in the protocol. Participants are expected to be in the study only for the time required to conduct the RHC and the Doppler echocardiographic study.

Exclusion Criteria

Exclusion criteria will include:

Severe pulmonary hypertension that is O2-dependent History of allergy to Optison® Hypersensitivity to perflutren, blood, blood products or albumin History of patent foramen ovale (PFO) or atrial septal defect (ASD) Known or suspected right-to-left, bi-directional, or transient right-to-left cardiac shunts Pregnancy Breastfeeding Advanced liver disease

Withdrawal Criteria

Withdrawal criteria will include:

Sustained ventricular arrhythmias at the time of the procedure Evidence of PFO or ASD at the time of the Doppler echocardiographic study Development of hypersensitivity or allergy to Optison®

Right Heart Catheterization

Invasive hemodynamic assessment by Swan-Ganz catheterization will be performed according to the standard protocol of the Cardiac Catheterization Laboratory. The following parameters will be recorded:

Right atrial pressure Right ventricular pressure Pulmonary artery pressure (PAP) Pulmonary capillary wedge pressure (PCWP) Cardiac output by thermodilution method (CO)

Pulmonary vascular resistance (PVR) will be calculated according to the following formula:

PVR=80*(Mean PAP-Mean PCWP)/CO

Blood Drawing During the right heart catheterization a total of 30 mL of blood will be drawn when the tip of the catheter is in the main pulmonary artery, in the right pulmonary artery, and in the wedged position. Blood will be collected in tubes, placed in ice and subsequently processed. Whole blood, serum and plasma will be frozen and stored for measurement of various biomarkers (e.g. osteoprotegerin and endothelin-1).

Doppler Echocardiographic Study Echocardiographic image acquisition will be performed using routine transthoracic echocardiography standards. Right ventricular outflow tract velocity-time integral (RVOT

VTI) will be measured. The tricuspid annular plane systolic excursion (TAPSE) will be assessed in the apical four chamber view with the M-mode cursor through the lateral tricuspid annulus. The peak velocity (v) of the tricuspid regurgitation jet will be measured by Doppler echocardiography in multiple projections, and the tricuspid pressure regurgitation gradient (P) will be calculated from the modified Bernoulli equation using the highest velocity obtained:

P=4v^2

The inferior vena cava will be visualized in the subcostal view throughout multiple respiratory cycles and IVC diameter will be measured at end expiration and end inspiration to assess right atrial pressure according to current criteria. The ratio of peak tricuspid regurgitation velocity (TRV) and RVOT VTI, which has been shown to correlate with PVR, will be calculated.

Monitoring The investigators will perform monitoring after the Optison® injection according to the package insert.

Statistical Analyses The primary analyses will aim to correlate noninvasive and invasive RAP or PASP measures. Secondary analyses will compare such measures by assessment modality. To address the first specific goal, Pearson's correlation coefficient will be estimated for RAP obtained noninvasively and by RHC. For the remaining three goals, the same approach will be utilized to correlate the outcome of interest measured noninvasively and by RHC. For example, in the second goal, Pearson's correlation coefficient will be estimated for PASP measured noninvasively by agitated saline solution administration and invasively via RHC. For each specific goal, measurements via the two modalities will be displayed graphically using scatterplots. To summarize the nature of this relationship, flexible regression methods, including smoothing splines regression, will be utilized in each specific goal. In secondary analyses, for each specific goal, comparisons of the two outcomes (RAP or PASP values) measured using the noninvasive and the invasive approaches will be made based on paired t-test, if the outcomes are normally distributed. Otherwise, Wilcoxon's signed rank test shall be employed. Detailed summaries of the RAP and PASP values obtained noninvasively or invasively will be presented for each specific goal. Summaries will include the mean, median, standard deviation, minimum and maximum values. Regression models will be explored to gain a better understanding of the underlying patterns in RAP or PASP values, while adjusting for important patient characteristics such as demographics. An overall type I error of 5% will be maintained. To ensure this, each of the aims will be allocated a 1.25% type I error. For each specific goal, a sample of 100 participants will yield statistical power in excess of 85% to detect a Pearson correlation level of ±0.35. To detect increased correlation levels of ±0.50 or more extreme, power exceeds 99%. Consequently, based on a sample of size 75, this study is well equipped to detect realistic level of correlation between RAP or PASP values obtained by noninvasive and invasive methods. Statistical significance for each of the four primary analyses will be performed at 1.25% alpha level. Significance level in all secondary and additional exploratory analyses will be set at 5%.

3. Anticipated Results The investigators expect to collect accurate estimates of the correlations between cardiac right-sided pressures assessed noninvasively by Doppler echocardiography and the gold standard RHC-measured pressures. Additionally, the investigators expect to demonstrate an improvement in the accuracy of Doppler echocardiography measurements with the use of an intravenous contrast agent. Finally, the investigators expect to find associations between biomarkers level and pressures measured during the right heart catheterization.

4. Potential Pitfalls Insufficient enrollment of research participants. Technical difficulty with echo images.

ELIGIBILITY:
Inclusion Criteria:

* Unselected consecutively patients 18 to 80 years old referred for RHC to the Cardiac Catheterization Laboratory of Northwestern Memorial Hospital. The informed consent for RHC will be obtained as part of the clinical assessment.

Exclusion Criteria:

* Severe pulmonary hypertension that is O2-dependent
* History of allergy to Optison®
* Hypersensitivity to perflutren, blood, blood products or albumin
* History of patent foramen ovale (PFO) or atrial septal defect (ASD)
* Known or suspected right-to-left, bi-directional, or transient right-to- left cardiac shunts
* Pregnancy
* Breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unselected consecutively patients 18 to 80 years old referred for RHC to the Cardiac Catheterization Laboratory of Northwestern Memorial Hospital.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Simultaneous Noninvasive and Invasive measurements of PA pressures | Data acquisition wll be obtained as soon as the RHC is performed, expected average of 5 weeks
  Doppler echo measurements:
  Estimated pulmonary artery (PA) systolic pressure without any contrast (units = mmHg) Estimated PA systolic pressure with agitated saline contrast (units = mmHg) Estimated PA systolic pressure with echocardiographic contrast (units = mmHg) Right heart catheterization (RHC) measurements: Invasively measured PA systolic pressure (units = mmHg)

SECONDARY OUTCOMES:
Simultaneous assessment of IVC collapsibility and invasive right atrial pressure measurement | Immediately will be noted as soon as PHC is performed, expected average of 5weeks
  Echo measurement: Assessment of inferior venacava diameter and collapsibility to assess RA pressure measurement (Units: diameter in cm, and non-invasive RAP in mm Hg) Right heart catheterization(RHC) measurement: Invasively measured right atrial pressure (units= mm Hg) The assessment of inferior diameter and collapsibility will allow determination of RA pressure non-invasively.

CONTACTS AND LOCATIONS:
Overall Officials: Kameswari Maganti, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Result] Galie N, Hoeper MM, Humbert M, Torbicki A, Vachiery JL, Barbera JA, Beghetti M, Corris P, Gaine S, Gibbs JS, Gomez-Sanchez MA, Jondeau G, Klepetko W, Opitz C, Peacock A, Rubin L, Zellweger M, Simonneau G; ESC Committee for Practice Guidelines (CPG). Guidelines for the diagnosis and treatment of pulmonary hypertension: the Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS), endorsed by the International Society of Heart and Lung Transplantation (ISHLT). Eur Heart J. 2009 Oct;30(20):2493-537. doi: 10.1093/eurheartj/ehp297. Epub 2009 Aug 27. No abstract available. PMID 19713419